CLINICAL TRIAL: NCT04201067
Title: Large-Scale Metabolomic Profiling for the Diagnosis of Inborn Errors of Metabolism
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, David R. Deyle, Principal Investigator, Mayo Clinic
Other Study IDs: 16-004682; U54NS115198-01 (NIH)
Record Dates: First submitted 2019-12-08; First posted 2019-12-17 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Congenital Disorders of Glycosylation
MeSH Terms: conditions — Congenital Disorders of Glycosylation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Stool, urine, DBS, fibroblasts, and blood can be retained for biomarker testing. DNA may be a part of this testing in the future.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Researchers are trying to determine the efficacy of a global metabolomic approach in testing for and diagnosing inborn errors of metabolism as opposed to traditional testing methods.

DETAILED DESCRIPTION:
Residual samples will be tested for a variety of biomarkers that may lead to better understanding of these disorders and help develop treatment options.

ELIGIBILITY:
Inclusion Criteria:

* All individuals with specimens in Biochemical Genetics Laboratory and from patients collected under another IRB who have agreed to share samples/data

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: These individuals will likely have a congenital disorder of glycosylation or other metabolic disease.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Quantify N-linked glycan intermediates in plasma and urine | length of study, up to 5 years
  Measure N-linked glycan intermediates in plasma and urine from PMM2-CDG patients.
Develop quantitative biomarkers for PGM1-CDG patients to monitor the efficacy of galactose therapy. | length of study, up to 5 years
  Measure the 41 plasma N-glycan levels in 9 PGM1-CDG patients before and after galactose therapy.
Develop quantitative biomarkers for SLC35A2-CDG patients and monitor galactose therapy efficacy. | length of study, up to 5 years
  Measure levels of plasma N-glycans from 10 SLC35A2-CDG patients before and after galactose therapy.
Validate biomarker to diagnose and follow NGLY1 deficiency and monitor N-acetylglucosamine (GlcNAc) therapy response. | length of study, up to 5 years
  Measure the level of Sia-Gal-GlcNAc-Asn biomarker excretion during GlCNAc therapy.
Validate novel diagnostic biomarkers for ALG13-CDG | length of study, up to 5 years
  Measure GlcNAc-β-Asn on glycoproteins in the cells from the already available fibroblast of 9 ALG13 patients.

CONTACTS AND LOCATIONS:
Overall Officials: David Deyle, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Information and samples can be shared at PI's discretion.
Supporting Information: Study Protocol
Time Frame: length of study

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials